CLINICAL TRIAL: NCT02169518
Title: Changes in Paraoxonase Activity, HDL Properties, Inflammatory Markers and Corneal Innervation in Post-bariatric Surgery Patients, Type 1 Diabetics With and Without Nephropathy, Type 2 Diabetics, and During an Oral Glucose Tolerance Test.
Brief Title: Paraoxonase and HDL Qualities in Glycaemia and Inflammation
Acronym: PON1
Status: Recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: British Heart Foundation (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PON2011
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus; Bariatric Surgery Candidate
Keywords: PON1 activity; HDL functionality; LDL oxidation; Diabetes Mellitus Type 1; Obesity; Diabetes Mellitus Type 2; Bariatric Surgery
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetes Arm: Patients with Type 1 and Type 2 diabetes
- Bariatric Arm: Obese patients scheduled for bariatric surgery

SUMMARY:
The incidence of coronary heart disease (CHD) is significant in the super-obese and diabetics.

Inflammation is believed to play an important part in the development of CHD, and the large collection of abdominal fat in the obese person is a vast source of inflammation. Diabetics have abnormal glucose and cholesterol metabolism which ultimately compromise their bodies' circulatory system and nerve function.

Cholesterol plays a vital role in CHD. Low-density lipoprotein (LDL) particles carry cholesterol and deposit it in blood vessel walls which become damaged as a result. When LDL particles undergo changes chemically (called oxidation) or as a result of high circulating blood glucose (called glycation), they become more harmful to the body. High-density lipoprotein (HDL) particles have a protective function in CHD. Not only do they transport cholesterol away from the blood vessels to the liver to be broken down, they have properties against oxidation and inflammation. These properties are related to the activity of an enzyme on HDL called paraoxonase 1(PON1).

Super-obese patients are increasingly treated by weight-reducing surgery (bariatric surgery). In this study we examine whether weight loss following bariatric surgery results in reduced inflammatory state, improved HDL function (higher PON1 activity), better control of blood glucose and less nerve damage.

We will study PON1 activity, inflammation and glucose control in patients with type 1 diabetes (with and without kidney damage) and type 2 diabetes. We will also study the effects of rapidly rising blood glucose levels on PON1 and glycated LDL in patients undergoing oral glucose tolerance test.

DETAILED DESCRIPTION:
High-density lipoprotein (HDL) is known to have a protective role in cardiovascular disease. Apart from transporting cholesterol from peripheral blood vessels back to the liver where it is processed, HDL has the ability to inhibit chemical changes (called oxidation) to low-density lipoprotein (LDL) which would make the latter more toxic to the body. HDL can also stop inflammatory particles from damaging the vessel walls. The anti-oxidation and anti-inflammatory properties of HDL are associated with an enzyme on HDL called paraoxonase 1 (PON1). It is not the level of measured HDL but the level of PON1 activity that is important in preventing cardiovascular disease. PON1 activity determines the quality of HDL and the effect against vascular disease.

Obese patients accumulate most of the fat within their abdomen (termed visceral fat). It is known that visceral fat produces large quantities of inflammatory particles so that obese patients have increased systemic inflammation and thus higher risk of vascular disease. The impact of heightened inflammatory status on HDL functions and PON1 activity is not known. Weight-reducing (bariatric) surgery can result in significant weight loss in obese patients. It is unclear whether the weight loss is associated with improvement in HDL functions, possible reversal of lipoprotein abnormalities and other physiological parameters. We plan to study a population of obese patients scheduled to have bariatric surgery before and after the surgery and compare the results with a matching population of healthy control patients.

Diabetic patients are at increased risk of developing cardiovascular disease. HDL in diabetic patients is often dysfunctional. Even though HDL levels are normal, PON1 activity may be reduced. LDL is able to interact with raised levels of blood glucose (called glycation) and become more harmful to the body. Glycation of lipoproteins associated with PON1 may affect PON1 activity. We plan to study glycated lipoproteins and PON1 activity in a population of diabetic patients who have either type 1 or type 2 diabetes. Some of the type 1 diabetics will have diabetic kidney disease, these patients are known to be particularly at high risk of cardiovascular complications. We also plan to recruit a cohort of patients who do not have diabetes but who have had an abnormal blood glucose test. These patients will be having an oral glucose tolerance test (OGTT) which establishes whether they have diabetes. During the OGTT, patients are given an oral glucose load which results in a rapid rise in blood glucose. We will see if this accelerated change in blood glucose level has any effects on the glycation of lipoproteins.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 diabetes who are not receiving lipid-lowering drugs, omega fatty acid supplements or thiazolidinediones and without clinical and/or ECG evidence of CHD.

Type 2 diabetic patients who are not receiving omega fatty acid supplements or thiazolidinediones and without clinical and/or ECG evidence of CHD.

Patients with impaired fasting glucose undergoing oral glucose tolerance test. Patients scheduled for bariatric surgery. Healthy controls who have no major acute or chronic illness, are not receiving regular medication and not taking omega fatty acid supplements, do not have clinically overt ischaemic heart disease.

Subjects (male and female) aged between 20 and 75. Subjects who have capacity and understanding for informed consent process.

Exclusion Criteria:

* Type 1 diabetics using lipid lowering therapy, thiazolidinediones, omega fatty acid supplements. History and/or ECG evidence of ST segment changes indicative of CHD.

Type 2 diabetics receiving thiazolidinediones, omega fatty acid supplements. History and/or ECG evidence of ST segment changes indicative of CHD.

Healthy controls who have any history of CHD, vascular insufficiency, or diabetes. Use of any lipid-lowering drug or omega fatty acid supplements.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 patients with type 1 diabetes 60 control subjects for type 1 diabetics 60 patients with type 2 diabetes 60 control subjects for type 2 diabetics 60 patients undergoing oral glucose tolerance test 120 patients scheduled for bariatric surgery - lipoprotein group 120 control subjects for bariatric patients 60 patients scheduled for bariatric surgery - nerve function & structure group
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-07-05 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Paraoxonase activity is measured using a semi-automated microtitre plate method. | 1 day
  Paraoxonase activity is measured and analysed in the groups of patients with defined medical conditions according to the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Handrean Soran, MD FRCP, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Central Manchester University Hospitals NHS Foundatioon Trust, Manchester, Lancashire, United Kingdom

REFERENCES:
- [Derived] Yadav R, Hama S, Liu Y, Siahmansur T, Schofield J, Syed AA, France M, Pemberton P, Adam S, Ho JH, Aghamohammadzadeh R, Dhage S, Donn R, Malik RA, New JP, Jeziorska M, Durrington P, Ammori BA, Soran H. Effect of Roux-en-Y Bariatric Surgery on Lipoproteins, Insulin Resistance, and Systemic and Vascular Inflammation in Obesity and Diabetes. Front Immunol. 2017 Nov 15;8:1512. doi: 10.3389/fimmu.2017.01512. eCollection 2017. PMID 29187850